CLINICAL TRIAL: NCT02490852
Title: Study of Nutritional Suitability of a New Infant Formula for Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ausnutria Hyproca B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AUS/015513
Record Dates: First submitted 2015-06-29; First posted 2015-07-07 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2018-11

CONDITIONS: Growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Investigational Infant formula (Experimental): Healthy term infants fed exclusively the investigational Infant Formula
  Interventions: Other: Investigational infant formula
- Commercially available Infant formula (Active Comparator): Healthy term infants fed exclusively a commercially available Infant Formula
  Interventions: Other: Active Comparator: Commercially available Infant formula
- Human milk (Active Comparator): Healthy term infants fed exclusively human milk
  Interventions: Other: Active Comparator: Human milk

INTERVENTIONS:
Other: Investigational infant formula — fed ad libitum
  Arms: Investigational Infant formula
Other: Active Comparator: Commercially available Infant formula — fed ad libitum
  Arms: Commercially available Infant formula
Other: Active Comparator: Human milk — fed ad libitum
  Arms: Human milk

SUMMARY:
This is a growth study of full-term infants. The growth of infants fed the investigational formula will be compared with infants fed a control formula. A breastfeeding arm will be used as reference.

ELIGIBILITY:
Inclusion Criteria:

* Healthy full term infant (37-42 weeks of gestational age)
* Birth weight 2,500 to 4,500 g
* Infant's mother willing and able to exclusively breast feed or infant's parent(s)/caregiver(s) willing to exclusively use randomized infant formula during study participation
* Parent(s)/caregiver(s) able to attend visits and willing to complete the subject diary
* Informed consent signed by parent(s)/caregiver(s)

Exclusion Criteria:

* Congenital illness or malformation that may affect infant feeding or normal growth
* Gastrointestinal disorders
* Suspected or known allergy to milk protein for formula groups
* Known food allergies in parents or siblings for formula groups
* Multiples
* Readmission to hospital for longer than 3 days for another reason than hyperbilirubinemia prior to enrollment
* Infant participating in another clinical study
* Infant's family unable to comply with the protocol according to the investigators's assessment

Max Age: 13 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2015-08; Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Weight gain | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Falco Panzer, Dr. Med., Principal Investigator — Kinderärztliche Gemeinschaftspraxis
Locations (18):
- Vienna, Austria
- Croatia (8):
  - Dubrovnik
  - Kutina
  - Split
  - Vukovar
  - Zadar
  - Zagreb
  - Zaprešić
  - Đakovo
- Germany (7):
  - Bramsche
  - Hamm
  - Herford
  - Mannheim
  - Mönchengladbach
  - Wesel
  - Wuppertal
- Spain (2):
  - Barcelona
  - Madrid